CLINICAL TRIAL: NCT00750113
Title: A Multicenter Study Evaluating the Efficacy of Nifedipine GITS - Telmisartan Combination in Blood Pressure Control and Beyond: Comparison of Two Treatment Strategies.
Brief Title: Study Evaluating the Efficacy of Nifedipine GITS - Telmisartan Combination in Blood Pressure Control.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12313; 2006-006436-22 (EudraCT Number)
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Nifidipine
- Arm 2 (Experimental)
  Interventions: Drug: Telmisartan
- Arm 3 (Experimental)
  Interventions: Drug: Nifedipine/Telmisartan

INTERVENTIONS:
Drug: Nifidipine — Tablets 20 Mg daily for 4 weeks then combination therapy
  Arms: Arm 1
Drug: Telmisartan — Tablets 80 Mg daily for 4 weeks then combination therapy
  Arms: Arm 2
Drug: Nifedipine/Telmisartan — 2 drugs (20 Mg Nifedipine/80 Mg Telmisartan) Combination therapy since the beginning
  Arms: Arm 3

SUMMARY:
Patients having uncontrolled or poorly controlled hypertension are at risk of experiencing cardiovascular events such as myocardial infarction or stroke. To reduce this risk an appropriate antihypertensive therapy should allow to reach a target blood pressure of less than 130/80 mmHg in order to maximise cardiovascular protection.The purpose of this study is to evaluate the efficacy in blood pressure control when anti-hypertensive therapy is initiated with a combination of low dose Nifedipine GITS and Telmisartan compared to a regimen starting with monotherapy before adding the other drug.The primary efficacy parameter will be the 24 hour mean systolic Blood Pressure on Ambulatory Blood Pressure Monitoring (ABPM) at 16 weeks of treatment compared to baseline

ELIGIBILITY:
Inclusion Criteria:

* Hypertension (office systolic blood pressure > 135 mmHg), untreated or poorly controlled but stable antihypertensive regimen for >/= 4 weeks
* Presence of type 2 diabetes mellitus or target organ damage (echocardiographic or electrocardiographic left ventricular hypertrophy or microalbuminuria)
* Presence of a metabolic syndrome, i.e at least two of the following [(from letter (a) to letter(d)] in patients with organ damage or at least one of the following [from letter (b) to letter (d)] in patients with diabetes mellitus: (a) impaired glucose tolerance (fasting plasma glucose 110 -125 mg/dl) (b )raised serum triglycerides (>/= 150 mg/dl) or comitant use of statins for this indication(c) low HDL cholesterol (males: < 40 mg/dl, females: < 50 mg/dl)(d) waist circumference >102 cm in men and >88 cm in women
* Age: 18-75 years
* Negative pregnancy test in females
* Written informed consent

Exclusion Criteria:

* Concomitant treatment with AT1-antagonists e.g. losartan, eprosartan, telmisartan) or calcium-antagonists (e.g. amlodipine, felodipine, isradipine, nifedipine, nimodipine).
* Concomitant treatment with any other antihypertensive medication that cannot be safely withdrawn at entry (i.e taken on a stable regimen for >/= 4 week) and that won't possibly be kept stable over the whole duration of the study.
* Concomitant treatment with known cytochrome P450-3A4 inhibitors (e.g cimetidine, anti-HIV protease inhibitors e.g. ritonavir, azole anti-mycotics eg. Ketoconazole, digoxin, quinidine, tacrolimus) or inducers such as anti-epileptic drugs (eg. phenytoin, carbamazepine and phenobarbitone) or rifampicin
* Concomitant treatment with potassium sparingdiuretics.
* Malignant, severe or labile essential hypertension, orthostatic hypotension
* Cardiovascular shock
* Evidence of secondary form of hypertension, including coarctation of the aorta, hyperaldosteronism, renal artery stenosis or pheochromocytoma
* Myocardial infarction or unstable angina within the previous 12 months
* Severe cardiac valve disease
* Severe rhythm or conduction disorder:
* Cerebrovascular ischaemic event (stroke, transient ischaemic attack) within the previous 12 months
* History of intra-cerebral haemorrhage or sub-arachnoid haemorrhage within the previous 12 months
* Type 1 diabetes mellitus
* Proteinuria (determined by uristix)
* BMI > 34
* Uncorrected hypokalemia or hyperkalemia, potassium outside the range 3.0 to 5.5 mmol/l
* Sodium depletion and/or hypovolemia
* Gastrointestinal disease resulting in the potential for malabsorption)
* Liver disease or transaminase (AST, ALT) levels > 3 x the upper limit of normal range.
* Renal failure, creatinine >2.0 mg/dl
* General Exclusion Criteria: any malignant disease that has required treatment within the last five years, dementia or psychosis, history of non-compliance, alcoholism or drug abuse, treatment with any other investigational drug in the 30 days prior to entering the study, pregnancy and lactation, known state of allergy or hypersensitivity to nifedipine or any other dihydropyridine or to telmisartan, any surgical or medical condition which at the discretion of the investigator place the subject at higher risk from his/her participation in the study or are likely to prevent the subject from complying with the requirements of the study or completing the trial period, history of non compliance to medical regimens or subjects unwilling to comply with the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter will be the 24 hour mean systolic Blood Pressure on Ambulatory Blood Pressure Monitoring (ABPM) | at 16 weeks of treatment compared to baseline

SECONDARY OUTCOMES:
Office blood pressure, response rate (> 10mmHg decrease control rate (< 130/80) mean SBP, mean DBP. | 8, 16 weeks of treatment
ABPM: % patients achieving BP < 125/80 mmHg morning BP increase/surge,24h mean diastolic BP,day average BP, night average BP,BP variability, pulse pressure through to peak ratio,smoothness index dipping or non dipping | 8, 16 and 24 weeks
Microalbuminuria in subgroup (any reduction) | 8, 16 and 24 weeks
Metabolic parameters: fasting blood glucose, total cholesterol, LDL cholesterol, HDL cholesterol, Triglycerides | 8, 16 and 24 weeks
Inflammatory markers: sRAGE (soluble receptors for advanced glycation end products) eotaxin-3, CRP (C-Reactive Protein) | 8, 16 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (39):
- Italy (28):
  - Pozzilli, Isernia
  - Monza, Monza-Brianza
  - Somma Lombardo, Varese
  - Ancona
  - Bologna
  - Brescia
  - Broni
  - Catania
  - Cinisello Balsamo
  - Ferrara
  - L’Aquila
  - Milan
  - Napoli
  - Novara
  - Padua
  - Palermo
  - Pavia
  - Perugia
  - Pisa
  - Reggio Emilia
  - Roma
  - Sassari
  - Siena
  - Syracuse
  - Treviso
  - Trieste
  - Varese
  - Venezia
- Spain (11):
  - Ferrol, A Coruña
  - Badajoz, Badajoz
  - Badalona, Barcelona
  - Ciudad Real, Ciudad Real
  - Jerez de la Frontera, Cádiz
  - Las Palmas de Gran Canaria, Las Palmas
  - Madrid, Madrid
  - Málaga, Málaga
  - Gijón, Principality of Asturias
  - Benigànim, Valencia
  - Valencia, Valencia

REFERENCES:
- [Result] Mancia G, Parati G, Bilo G, Choi J, Kilama MO, Ruilope LM; TALENT investigators. Blood pressure control by the nifedipine GITS-telmisartan combination in patients at high cardiovascular risk: the TALENT study. J Hypertens. 2011 Mar;29(3):600-9. doi: 10.1097/HJH.0b013e328342ef04. PMID 21252701
- See also: Click here and search for Bayer Product infromation provided by EMA — http://www.clinicaltrialsregister.eu